CLINICAL TRIAL: NCT05183581
Title: Feeling Hot 1: Investigating the Influence of Clothing and Blankets on Penile Skin Temperature During Male Sexual Arousal
Brief Title: Feeling Hot 1: Environmental Influences of Overnight Measurement on Skin Temperature of the Erectile Penis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Antonius Hospital (Other)
Responsible Party: Principal Investigator, Hille Torenvlied, Coordinating Investigator, St. Antonius Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 79920
Record Dates: First submitted 2021-12-22; First posted 2022-01-10 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Erectile Dysfunction
Keywords: Erectile Dysfunction; RigiScan; Nocturnal erection; Penile temperature
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Visually aroused erection (naked, clothing, blankets) (Other): Randomisation of the order of visually aroused erection will be conducted:
  1. Naked - Naked & Blanket - Clothing & Blanket
  2. Naked - Clothing & Blanket - Naked & Blanket
  3. Naked & Blanket - Naked - Clothing & Blanket
  4. Naked & Blanket - Clothing & Blanket - Naked
  5. Clothing & Blanket - Naked - Naked & Blanket
  6. Clothing & Blanket - Naked & Blanket - Naked
  Interventions: Device: Feeling Hot sensor system

INTERVENTIONS:
Device: Feeling Hot sensor system — The Feeling Hot sensor system consists of two temperature probes placed on the penis and outer thigh of the test subject to measure skin temperature during erection.

SUMMARY:
The Feeling Hot studies focus on the proof-of-principle of using temperature sensing as a tool to detect nocturnal erections. In the Feeling Hot 1 study the influence of environmental factors of overnight measurements are studied in a controlled setting. Healthy individuals will have visually aroused erections in different circumstances (naked, clothing, blankets) to determine the feasibility of this new measurement method for nocturnal erection detection in the search to modernize erectile dysfunction diagnostics.

DETAILED DESCRIPTION:
Differentiation in nature of erectile dysfunction (ED) is currently made by nocturnal erection detection with the RigiScan. The RigiScan uses outdated software, measurements are user unfriendly and system components are out of stock. In the search of modernizing erectile dysfunctions diagnostics, the question has arisen whether temperature measurements can function as a tool for nocturnal erection detection. With the absence of a pressure component, the patient experience should improve. Literature and mathematical modelling studies have shown that the penile temperature increases significantly during erection. However, it is unclear what the influence of environmental factors such as blankets and clothing is on the increase in penile temperature during erection. The Feeling Hot 1 study explores the effects of these environmental factors in a controlled setting to gain insight into the possibility of using temperature sensing to detect nocturnal erections.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Aged 18 - 29 years
* Capable of getting visually arousable erections

Exclusion Criteria:

* Test subject unwilling to sign informed consent
* Test subject with erectile dysfunction
* IIEF-5 score below 17
* Medical history consisting of sickle cell anaemia, atherosclerosis and/or diabetes type I/II

Ages: 18 Years to 29 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2022-05-17 (Actual); Primary Completion 2022-06-09 (Actual); Study Completion 2022-07-27 (Actual)

PRIMARY OUTCOMES:
Temperature increase | 10 minutes
  Increase in penile skin temperature during erection
(De)tumescence duration | 10 minutes
  Duration of increased penile skin temperature during erection

SECONDARY OUTCOMES:
Difference between sexual and nocturnal erections | 10 hours
  Penile and outer thigh temperature increase difference between sexual and nocturnal erection

CONTACTS AND LOCATIONS:
Overall Officials: Jack Beck, Dr.,MD., Principal Investigator — Urologist, St. Antonius Ziekenhuis
Locations (1):
- St. Antonius Ziekenhuis, Nieuwegein, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No